CLINICAL TRIAL: NCT06019195
Title: Time Restricted Eating for Prevention of Age-related Vascular Cognitive Decline in Older Adults
Brief Title: The Effect of Intermittent Fasting on Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16102; 1R21AG080775-01A1 (NIH)
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Intermittent Fasting; Aging
Keywords: Intermittent Fasting; Aging
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time restricted eating (Experimental): not more than 10 hrs. eating window daily goal for 6 months
  Interventions: Other: Time restricted eating

INTERVENTIONS:
Other: Time restricted eating — not more than 10 hrs. eating window daily goal for 6 months
  Other Names: intermittent fasting

SUMMARY:
The central hypothesis of this study is that closer adherence to time restricted eating (TRE) will improve endothelial function, neurovascular (NVC) responses, resulting in improved cognitive performance, potentially through activation of SIRT1-dependent vasoprotective pathways.

DETAILED DESCRIPTION:
This hypothesis will be tested by assessing the effect of TRE (not more than 10hr eating window each day for 6 months) in healthy older adults (55-80 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55 and ≤80 years of age
* Adequate hearing and visual acuity to participate in the examinations
* Ability to read and write in English
* Competence to provide informed consent.
* Mini Montreal Cognitive Assessment ≥12
* Mini Nutritional Assessment ≥12

Exclusion Criteria:

* Vision or hearing impairment that would impair the ability to complete study assessments
* Active CNS disease including multiple sclerosis, uncontrolled seizures, active brain cancer
* Cerebrovascular accident other than TIA within 60 days prior to Visit 0
* Major psychiatric disease, including major depression not currently controlled on medications, alcohol or drug abuse
* Diabetics prescribed sulfonylureas, meglitinides, and insulin
* Any other medical condition which, in the opinion of investigator, would render the patient inappropriate or too unstable to complete the study protocol

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Change in neurovascular coupling using functional near infrared spectroscopy (fNIRS) | baseline, up to 6 months
  Functional near infrared spectroscopy (fNIRS) will be performed during the cognitive n-back task. fNIRS approach generates data that represent a relative change in oxygenated and deoxygenated hemoglobin measured over the cortical brain tissues. Neurovascular coupling will be evaluated as a change in oxy- and deoxy-hemoglobin between before and after completion of study.
Change in neurovascular coupling using the dynamic retinal vessel analysis | baseline, up to 6 months
  Flicker light-induced dilation of the retinal vessels (percentage increase over baseline diameter) will be measured in the right or left eye of each study participant using the Dynamic Vessel Analyzer (DVA, IMEDOS Systems, Jena, Germany). The change in retinal vessel diameters is tracked and reported as a %change from baseline, before and after completion of study.
Change in EEG spectra | baseline, up to 6 months
  EEG signal will be collected to generate spectral data. These data will be used for comparison of EEG activity between before and after treatment. Units of measure - power spectral density. Reported as a %change from baseline, before and after completion of study.

SECONDARY OUTCOMES:
Change in microvascular endothelial function | baseline, up to 6 months
  Changes in microvascular endothelial function will be assessed using laser speckle contrast imaging (LSCI) in the hand using the flow mediated dilation approach. The change in skin perfusion is calculated and reported as a %change from baseline, between before and after completion of study.
Change in arterial stiffness | baseline, up to 6 months
  The arterial stiffness will be measured using the pulse wave analysis approach (SphygmoCor, Atcor medical, Itasca IL, or similar). Analysis generated the augmentation index which will be used for comparison before and after completion of study.
Change in Glycocalyx - perfused boundary region | baseline, up to 6 months
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include perfused boundary region (um), and will be used for comparison before and after completion of study.
Change in capillary density | baseline, up to 6 months
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include capillary density (mm/mm^2), and will be used for comparison before and after completion of study.
Change in red blood cell velocity | baseline, up to 6 months
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include red blood cell velocity (um/sec), and will be used for comparison before and after treatment.
Change in Attention | baseline, up to 6 months
  The allocation of one's limited capacities to deal with an abundance of environmental stimulation will be measured in a combined "Flanker Inhibitory Control and Attention Test".Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline.
Change in Working Memory | baseline, up to 6 months
  The ability to store information until the amount of information to be stored exceeds one's capacity to hold that information will be measured using the "List Sorting Working Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline.
Change in Executive Function | baseline, up to 6 months
  The capacity to plan, organize and monitor the executive of behaviors that are strategically directed in a goal-oriented manner will be measured using the "Dimensional Change Card Sort Test". Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline.
Change in Processing Speed | baseline, up to 6 months
  Pattern Comparison Processing Speed Test assesses the amount of information that can be processed within a certain unit of time. Items are simple so as to purely measure processing speed. Units of measure - score (from 0 to 130, bigger number is better). Reported as a %change from baseline.
Body composition | baseline, up to 6 months
  Weight and body composition using a bioimpedance scale and/or DXA scan. Reported as a %change from baseline, before and after completion of study
Dietary intakes | baseline, up to 6 months
  Dietary intake data for 24-hour recalls will be collected and analyzed using the Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool, version 2022, developed by the National Cancer Institute (https://epi.grants.cancer.gov/asa24). Estimated dietary intakes will be used to determine whether a participant was in a hypocaloric, eucaloric, or hypercaloric state during the intervention.
Total daily energy expenditure | baseline, up to 6 months
  Total daily energy expenditure will be estimated using the Mifflin-St. Jeor equation. Estimated total daily energy expenditure will be used to determine whether a participant was in a hypocaloric, eucaloric, or hypercaloric state during the intervention.
Change in blood metabolic panel markers | baseline, up to 6 months
  Complete metabolic panel. Reported as a %change from baseline, before and after completion of study
Change in Episodic Memory | baseline, up to 6 months
  Cognitive processes involved in the acquisition, storage and retrieval of new information, will be measured using the "Picture Sequence Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline.
Change in Language | baseline, up to 6 months
  Picture Vocabulary Test measures receptive vocabulary administered in a computer-adaptive test (CAT) format. Respondents select the picture that most closely matches the meaning of the word, before and after treatment. Unit of measure - overall score (bigger number is better). Reported as a %change from baseline.
Change in BOLD signal | baseline, up to 6 months
  Using fMRI, we will determine the changes in BOLD activation during standardized cognitive task. Reported as change in BOLD signal before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Andriy Yabluchanskiy, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Translational GeroScience Laboratory, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided
unidentified data may be shared via research repositories

REFERENCES:
- [Background] da C Pinaffi-Langley AC, Szarvas Z, Peterfi A, Kaposzta Z, Mukli P, Shahriari A, Muranyi M, Pinto CB, Owens CD, Adams C, Karfonta B, Rohan M, Tarantini S, Yabluchanskiy A. Time-restricted eating for prevention of age-related vascular cognitive decline in older adults: A protocol for a single-arm open-label interventional trial. PLoS One. 2024 Dec 9;19(12):e0314871. doi: 10.1371/journal.pone.0314871. eCollection 2024. PMID 39652561
- [Background] da C Pinaffi-Langley AC, Pinto CB, Mukli P, Peterfi A, Kaposzta Z, Owens CD, Szarvas Z, Muranyi M, Adams C, Shahriari A, Balasubramanian P, Ungvari Z, Csiszar A, Conley S, Hord NG, Anderson L, Tarantini S, Yabluchanskiy A. Energy metabolism dysregulation, cerebrovascular aging, and time-restricted eating: Current evidence and proof-of-concept findings. PNAS Nexus. 2024 Nov 8;3(11):pgae505. doi: 10.1093/pnasnexus/pgae505. eCollection 2024 Nov. PMID 39584020